CLINICAL TRIAL: NCT02488889
Title: Effects of Varenicline in Heavy Drinking Smokers
Acronym: VAR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution prior to enrollment of study participants
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23FT-0102
Record Dates: First submitted 2015-02-03; First posted 2015-07-02 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Cigarette Smoking; Alcohol Consumption
Keywords: Chantix
MeSH Terms: conditions — Cigarette Smoking; Alcohol Drinking | interventions — Varenicline; Ethanol; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline vs placebo (Active Comparator): Participants will be titrated on varenicline as follows: days 1-3, .5 mg per day; days 4-7, .5 mg twice per day, and days 7-12, 1 mg twice per day. Placebo and varenicline pills will be matched in number of pills and packaging of active medications.
  Interventions: Drug: Varenicline; Drug: Placebo pill (for varenicline)
- Alcohol beverage vs. placebo beverage (Active Comparator): During each experimental session, participants will ingest a beverage containing placebo (0.0 g/kg; 1% volume of ethanol as taste mask) or alcohol (0.8 g/kg). The beverage will be administered in clear plastic-lidded cups in 2 equal portions that will be consumed during a 5-minute interval and separated by a 5-minute interim rest. The beverages will contain 190-proof ethanol prepared with water, flavored drink mix, and a sucralose-based sugar substitute. Doses for women will be 85% of those of men to adjust for sex differences in total body water.
  Interventions: Drug: Alcohol; Drug: placebo beverage (for alcohol)

INTERVENTIONS:
Drug: Varenicline
  Arms: Varenicline vs placebo
Drug: Placebo pill (for varenicline)
  Arms: Varenicline vs placebo
Drug: Alcohol
  Arms: Alcohol beverage vs. placebo beverage
Drug: placebo beverage (for alcohol)
  Arms: Alcohol beverage vs. placebo beverage

SUMMARY:
This laboratory study will examine if varenicline can reduce alcohol-induced smoking lapse in heavy drinking smokers.

DETAILED DESCRIPTION:
There is a strong positive association between cigarette smoking and alcohol use both at the epidemiologic and behavioral levels. This co-use can create substantial impediments in smoking cessation. Approximately 25% of current smokers are heavy drinkers. Alcohol use is a risk factor for relapse during smoking cessation and is associated with lower odds of quitting smoking. Smokers are five times as likely to experience a smoking lapse during drinking episodes than at other times. Further, heavy drinking smokers experience more health consequences than individuals who are either only smokers or heavy drinkers, such as impairments in brain morphology and function and greater risk for various cancers. Given the high co-occurrence of smoking and drinking and the health risks associated with the co-use of these substances, it has been convincingly argued that heavy drinking smokers constitute a distinct sub-population of smokers with a unique clinical profile and treatment needs. Yet, there are no available pharmacological treatments or guidelines tailored to heavy drinking smokers, despite the evidence that this is a treatment-resistant sub-group. Thus, treatment development for heavy drinking smokers represents a highly significant and understudied research area. Varenicline is a first-line treatment for nicotine dependence that may also be effective in reducing alcohol use. Recent studies have indicated that varenicline reduces the pleasurable effects of alcohol and its self-administration in the laboratory, as well as alcohol craving and consumption in clinical trials. These findings suggest that varenicline is a promising medication for smoking cessation in heavy drinking smokers, as reducing alcohol craving and consumption may be a key component to effectively reducing smoking and preventing relapse in this sub-group.

In early abstinence, one of the most reliable predictors of relapse is the occurrence of a single smoking lapse, which is generally defined as smoking at least a puff of a cigarette. As much as 95% of smokers who experience a lapse will progress to relapse, which has led to the first lapse being theorized to represent the transition from abstinence to regular smoking. Alcohol consumption is one of the most consistently identified risk factors for a smoking lapse and, therefore, may contribute to the maintenance of nicotine dependence in heavy drinking smokers. Recent clinical trial and laboratory evidence suggests that varenicline is effective in reducing general smoking lapse behavior, although it is unknown whether this effect translates to alcohol-mediated smoking lapse behavior.

To address this important gap in the literature, this human laboratory study will use two laboratory paradigms, namely alcohol administration and a smoking lapse task, to examine clinically-relevant effects of varenicline among heavy-drinking smokers (i.e., individuals who smoke ≥ 10 cigarettes/day and who meet National Institute on Alcohol Abuse and Alcoholism (NIAAA) guidelines for heavy drinking). The investigators will enroll 22 non-treatment seeking heavy drinking smokers in a randomized, double-blind, placebo-controlled, crossover laboratory study, testing the efficacy of varenicline in reducing smoking behavior after controlled alcohol administration among heavy drinking smokers. All participants will be daily smokers (≥ 10 cig/day) who are also heavy drinkers according to NIAAA guidelines. Interested individuals will come in to the laboratory for an in-person screening visit and physical exam. Eligible participants will then be randomized to a medication sequence, varenicline (1 mg twice daily) or placebo. Medication will be titrated over a 12-day period and within each medication condition participants will complete two laboratory sessions on days 9 and 12. The laboratory sessions will consist of placebo-controlled alcohol administration followed by the McKee smoking lapse task. After completing both laboratory sessions for the first medication condition, and after a seven-day wash-out period, participants will be begin the second medication condition and again complete laboratory sessions on days 9 and 12 of the titration period (i.e., each participant will complete four laboratory sessions and experience all four combinations of varenicline/placebo pill and alcohol/placebo beverage). In each laboratory session, participants will receive a dose of alcohol [target breath alcohol concentration (BrAC) = 0.08 g/dl] or placebo beverage, in a randomized and double-blind fashion, and will then complete a smoking lapse task. In this paradigm, participants are presented with their preferred brand of cigarettes, a lighter, and an ashtray. Participants are then informed that they can begin a cigarette self-administration session or delay smoking in exchange for a fixed amount of monetary reinforcement. If the participant decides to smoke, they then begin the self-administration session in which they are again given the choice to smoke their preferred brand of cigarettes or receive a fixed monetary reinforcement for each cigarette that is not smoked. In addition to these smoking outcomes, measures of craving, mood, and subjective effects will be administered at baseline, after alcohol administration, and during the lapse paradigm. The study design allows for a within-subjects comparison of the effects of varenicline (versus placebo), alcohol (versus placebo), and their interaction on smoking behavior in the laboratory.

The Specific Aims of this project proposal are: Aim 1: To test whether varenicline is effective at reducing alcohol and cigarette craving, as well as reducing the acute subjective effects of alcohol and cigarettes; Aim 2: To test whether varenicline is effective at mitigating alcohol's effects on smoking lapse behavior; Aim 3: To test whether acute subjective response to alcohol is predictive of subsequent smoking lapse behavior and to examine if varenicline reduces this effect. The investigators hypothesize that varenicline, compared to placebo, will reduce cigarette and alcohol craving, attenuate subjective response to alcohol and cigarette smoking, and improve performance on the smoking lapse task by increasing the participant's ability to resist smoking. Furthermore, the investigators hypothesize that varenicline's ability to reduce alcohol craving and subjective response to an acute dose of alcohol will be directly predictive of performance on the smoking lapse task. Since heavy drinking smokers have been shown to be relatively treatment-resistant, the results of the current study could have sizable implications for supporting varenicline as a potential tailored treatment for this sizable and at-risk sub-group.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 21 and 55 and provide informed consent;
2. Smoke > 10 cigarettes per day for > 2 years and have a carbon monoxide (CO) > 10 ppm;
3. Report an interest in quitting smoking in the near future, but currently not in the process of quitting;
4. Report current heavy drinking according to NIAAA guidelines (62): for men, > 14 drinks per week or ≥ 5 drinks per occasion at least once per month over the past 12 months; for women, > 7 drinks per week or ≥ 4 drinks per occasion at least once per month over the past 12 months;
5. Not seeking or receiving treatment for alcohol use;
6. No current (last 12 months) diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V);
7. Negative urine toxicology screen for narcotics, amphetamines, and sedative hypnotics at screening;
8. No lifetime history of psychotic disorders, bipolar disorders, or major depression with suicidal ideation;
9. No current symptoms of moderate depression or higher, indexed by a score ≥ 20 on the Beck Depression Inventory-II (BDI);
10. No serious alcohol withdrawal symptoms as indicated by a score < 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised;
11. Not pregnant, nursing, or planning on becoming pregnant in the next month (if female);
12. Have no medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes);
13. Within normal limit aspartate transaminase (AST), alanine transaminase (ALT), or gamma-glutamyl transferase (GGT) levels;
14. Not currently on prescription medication that contraindicates use of VAR.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07-17 (Actual); Study Completion 2016-07-17 (Actual)

PRIMARY OUTCOMES:
The latency to initiate smoking during the delay period. Performance on the smoking lapse task | The task will begin five minutes after consumption of the alcohol or placebo beverage and last between 60 and 120 minutes based on performance
  In this task, eight cigarettes of the participants' preferred brand are placed in front of them with a lighter and an ashtray. Then, over the next 50 minutes they have the option to initiate a cigarette self-administration session at any point or delay initiation in exchange for monetary reinforcement. Once participants choose to end the delay period in order to smoke or resist smoking for the entire 50-minute delay period, they then participate in a 60-minute cigarette self-administration session, in which they are again given the choice to either smoke their preferred brand of cigarettes or receive monetary reinforcement for cigarettes not smoked. One primary outcome measure from this task is the latency to initiate smoking during the delay period.
The number of cigarettes smoked during the self-administration period. Performance on the smoking lapse task | The task will begin five minutes after consumption of the alcohol or placebo beverage and last between 60 and 120 minutes based on performance
  In this task, eight cigarettes of the participants' preferred brand are placed in front of them with a lighter and an ashtray. Then, over the next 50 minutes they have the option to initiate a cigarette self-administration session at any point or delay initiation in exchange for monetary reinforcement. Once participants choose to end the delay period in order to smoke or resist smoking for the entire 50-minute delay period, they then participate in a 60-minute cigarette self-administration session, in which they are again given the choice to either smoke their preferred brand of cigarettes or receive monetary reinforcement for cigarettes not smoked. The second primary outcome measure from this task is the number of cigarettes smoked during the self-administration period.

SECONDARY OUTCOMES:
Subjective effects of alcohol as measured by the Biphasic Alcohol Effects Scale (BAES) | up to 50- minutes of the delay period and 60-minutes of the self-administration session
Subjective effects of smoking as measured by the Nicotine Reward Scale (NRS) | up to 50- minutes of the delay period and 60-minutes of the self-administration session
The Drug Effects Questionnaire (DEQ) | up to 50- minutes of the delay period and 60-minutes of the self-administration session
Brief Questionnaire of Smoking Urges (B-QSU) | up to 50- minutes of the delay period and 60-minutes of the self-administration session

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States